CLINICAL TRIAL: NCT03478592
Title: Assessment of the New Automated Vitrification System "GAVI" for Early Cleaved Embryos Cryopreservation
Acronym: GAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/16/8766
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Fertility Disorders
Keywords: Slow-freezing; Vitrification; Automated system; Embryos; Implantation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reference technique slow freezing (Experimental): In reference technique slow freezing arm, embryon will be frozen with the conventional slow freezing procedure with the Freezal device apply a slow decreasing in temperature with moderate cryoprotector concentration
  Interventions: Other: reference technique
- vitrification technique (Experimental): In vitrification technique arm, embryon will be frozen with automated vitrification system
  Interventions: Other: vitrification technique

INTERVENTIONS:
Other: reference technique — Slow-freezing procedure is the reference technique, actually use at the Toulouse hospital, to cryopreserve embryos. Embryon are frozen with a slow freezing.
  Arms: reference technique slow freezing
Other: vitrification technique — Vitrification is the new technique to freeze embryons. In this study, the GAVI system will be use for for embryos automatically vitrification
  Arms: vitrification technique

SUMMARY:
The meta-analysis comparing the cryopreservation of human embryos by vitrification or slow-freezing suggested that more well design studies as randomized trials are necessary to identify the most successful method for cryopreservation. The efficacy of the vitrification with the GAVI system will be compared with the conventional slow freezing method through a randomized control trial. Couples in IVF attempt will be randomized at the day of embryo cryopreservation by the biologist. Supernumerary frozen embryos will be thawed and transferred in utero in case of failure of the "fresh" embryo transfer. The outcomes of the thawing and frozen/thawed embryo transfer will be assessed. In the two groups, the patients will benefit of the standard IVF procedures applied in the Assisted Reproductive Technologies (ART) center of Toulouse.

DETAILED DESCRIPTION:
The last decade has seen a development of a new cryopreservation technique called vitrification. Despite a lack of randomized control trials comparing slow-freezing and vitrification, vitrification seems to show better recovery rates and pregnancy outcomes. However vitrification is a manual, labour-intensive and highly skilled procedure, results can vary between embryologists and clinics. The GAVI system, an automation instrument with a novel closed system device has been developed. The present study would like to assess the outcomes for embryos automatically vitrification processed with the GAVI system compared with those processed with conventional reference technique of slow freezing.

The meta-analysis comparing the cryopreservation of human embryos by vitrification or slow-freezing suggested that more well design studies as randomized trials are necessary to identify the most successful method for cryopreservation. The efficacy of the vitrification with the GAVI system will be compared with the conventional slow freezing method through a randomized control trial. Couples in IVF attempt will be randomized at the day of embryo cryopreservation by the biologist. Supernumerary frozen embryos will be thawed and transferred in utero in case of failure of the "fresh" embryo transfer. The outcomes of the thawing and frozen/thawed embryo transfer will be assessed. In the two groups, the patients will benefit of the standard IVF procedures applied in the Assisted Reproductive Technologies center of Toulouse.

ELIGIBILITY:
Inclusion Criteria:

* Couple whose age is > 18 years and who are included in a IVF procedure with the possibility to cryopreserve embryos according to criteria applied at the hospital of Toulouse
* Signed informed consent by both partners in a couple
* Affiliation to a social security scheme for both partners of the couple

Exclusion Criteria:

* Couples who does not meet current requirements described by the bioethics law for accession to the ART procedure
* Positive plasma viral load for HIV, hepatitis C virus or hepatitis B virus during the year before the inclusion in one of the couple.
* One of the two partners (or both) is (are) in safeguarding justice, under guardianship or trusteeship.
* Couple included in another interventional study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Implantation rate of frozen/thawed embryos | 1 month
  The number of implantation embryo with cardiac activity in reference technique and in vitrification technic

SECONDARY OUTCOMES:
Percentage of intact blastomeres after thawing | 1 month
  It will be measured by microscopic evaluation by a biologist or an IVF laboratory technician at the time of thawing, routine very simple laboratory to do because at this early embryonic stage there are few cells: 4 to 8 cells and they are well individualized.
Implantation rate of transferred embryos. | 1 month
  number of implantation of transferred embryos in both technique
Live birth rates | 9 months after the implantation
  Number of live birth for reference technique and for vitrification technique

CONTACTS AND LOCATIONS:
Overall Officials: Roger Léandri, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hospital university of Toulouse, Toulouse, France